CLINICAL TRIAL: NCT01730846
Title: Does Doxazosin Attenuate Stress-induced Smoking and Improve Clinical Outcomes?
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Sherry McKee, Associate Professor of Psychiatry, Yale University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 1111009293; R21DA033597 (NIH)
Record Dates: First submitted 2012-11-09; First posted 2012-11-21 (Estimated); Results first posted 2017-12-20 (Actual); Last update posted 2018-02-20 (Actual); Status verified 2018-01

CONDITIONS: Smoking
Keywords: smoking lapse behavior; smoking cessation; doxazosin; medication effect on smoking lapse behavior; medication effect on smoking cessation; stress
MeSH Terms: conditions — Smoking; Smoking Cessation | interventions — Doxazosin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Doxazosin 4mg/day (Experimental): doxazosin 4mg/day
  Interventions: Drug: Doxazosin 4mg/day
- Placebo (Placebo Comparator): placebo control
  Interventions: Drug: Placebo
- Doxazosin 8mg/day (Experimental): doxazosin 8mg/day
  Interventions: Drug: Doxazosin 8mg/day

INTERVENTIONS:
Drug: Doxazosin 4mg/day — 4 mg/day with 3-week lead-in medication period. Maintained at steady state for duration of the study. 5-day taper at the end of the study.
  Other Names: Cardura
  Arms: Doxazosin 4mg/day
Drug: Placebo — Placebo
  Arms: Placebo
Drug: Doxazosin 8mg/day — 8 mg/day with 3-week lead-in medication period. Maintained at steady state for duration of the study. 5-day taper at the end of the study.
  Other Names: Cardura
  Arms: Doxazosin 8mg/day

SUMMARY:
The purpose of this study is to examine whether doxazosin will attenuate the ability of stress to precipitate smoking lapse behavior in treatment seeking daily smokers. Participants will participate in a smoking cessation attempt after the laboratory sessions.

ELIGIBILITY:
Inclusion Criteria:

* Ages 18-60
* Able to read and write English
* Smoker
* Motivated to Quit Smoking

Exclusion Criteria:

* Any significant current medical conditions that would contraindicate smoking
* Current Diagnostic and Statistical Manual of Mental Disorders (DSM-IV) abuse or dependence of other substances, other than nicotine dependence or alcohol abuse
* Positive test results at intake appointment on urine drug screens for illicit drugs
* Past 30 day use of psychoactive drugs including anxiolytics and antidepressants
* Women who are pregnant or nursing
* Suicidal, homicidal or evidence of current severe mental illness such as schizophrenia, bipolar disorder or major depression, or anxiety disorders
* Participants who have donated blood within the past 6 weeks
* Individuals who are currently taking other medications prescribed for smoking cessation
* Specific exclusions for administration of doxazosin or any alpha blocker

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 35 (Actual)
Dates: Start 2013-02; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sherry A McKee, PhD, Principal Investigator — Yale University
Locations (1):
- Yale Center for Clinical Investigations, Yale University, New Haven, Connecticut, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Placebo
  Placebo controlled
- 4mg/Day: doxazosin 4mg/day
  Doxazosin: 4 mg/day with 3-week lead-in medication period. Maintained at steady state for duration of the study. 5-day taper at the end of the study.
- 8mg/Day: doxazosin 8mg/day
  Doxazosin: 8 mg/day with 3-week lead-in medication period. Maintained at steady state for duration of the study. 5-day taper at the end of the study.
Period: Overall Study
Arm/Group | Placebo | 4mg/Day | 8mg/Day
Started | 11 | 11 | 13
Completed | 11 | 11 | 13
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | 4mg/Day | 8mg/Day | Total
Number analyzed (Participants) | 11 | 11 | 13 | 35
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.36 (9.29) | 34.82 (10.85) | 34.23 (9.83) | 35.40 (9.80)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 4 | 4 | 11
  Male | 8 | 7 | 9 | 24
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  African American | 5 | 1 | 7 | 13
  White | 6 | 6 | 4 | 16
  Hispanic | 0 | 2 | 1 | 3
  Other | 0 | 2 | 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: Latency (Min) to Initiate Ad-lib Smoking Session
Description: Latency to start smoking in the stress and neutral ad-lib smoking lab sessions. Subjects had the opportunity to delay smoking for 50 minutes (delay period). Once the subject decides to smoke, the 1 hour ad-lib smoking session begins. They can chose to smoke as little or as much as they wish.
Time Frame: 0 up to 50 minutes (Delay Period)
Measure: Mean (Standard Error); unit: minutes
Arm/Group | Placebo | 4mg/Day | 8mg/Day
Number analyzed (Participants) | 11 | 11 | 13
minutes
  Stress | 11.304 (7.407) | 32.128 (7.494) | 27.557 (6.409)
  Neutral | 23.474 (8.312) | 26.790 (8.410) | 23.776 (7.192)

2. Secondary Outcome: Number of Cigarettes Smoked During Ad-lib Session
Description: Number of cigarettes smoked during the stress and neutral ad-lib smoking period.
  Once the subject decides to smoke (delay period), the 1 hour ad-lib smoking period begins. They can chose to smoke as little or as much as they wish.
Time Frame: 60 minutes (ad-lib smoking period)
Measure: Mean (Standard Error); unit: number of cigarettes
Arm/Group | Placebo | 4mg/Day | 8mg/Day
Number analyzed (Participants) | 11 | 11 | 13
number of cigarettes
  Stress | 3.331 (0.563) | 1.890 (0.561) | 1.813 (0.493)
  Neutral | 2.139 (0.397) | 1.866 (0.396) | 1.688 (0.348)

ADVERSE EVENTS:
Time Frame: Titration period (3 weeks)
Description: Adverse events were assessed twice weekly with a symptom list during the 3-week titration period
Arm/Group | Placebo | 4mg/Day | 8mg/Day
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/11 | 0/13
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/11 | 0/13
Other Adverse Events (participants affected / at risk) | 4/11 | 6/11 | 7/13
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=11) | 4mg/Day (N=11) | 8mg/Day (N=13)
Fatigue (General disorders) | 0 | 2 | 4
Headache (General disorders) | 3 | 3 | 5
Dizziness (General disorders) | 0 | 3 | 2
Drowsiness (General disorders) | 0 | 5 | 3
Back pain (General disorders) | 0 | 1 | 0
Chest pain (Cardiac disorders) | 1 | 0 | 0
Pain (General disorders) | 0 | 0 | 1
Fast heartbeat (Cardiac disorders) | 0 | 1 | 3
Dry mouth (General disorders) | 1 | 3 | 1
Abnormal vision (General disorders) | 0 | 0 | 2
Impotence (General disorders) | 0 | 1 | 0
Urinary tract infection (General disorders) | 0 | 0 | 0
Increased sweating (General disorders) | 0 | 0 | 0
Anxiety (General disorders) | 0 | 1 | 0
Insomnia (General disorders) | 1 | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No